CLINICAL TRIAL: NCT03877341
Title: Sagittal Parameters After Mono Segmental Lumber Fusion: Interbody Versus Postrolateral Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fady Samy saeed, resident assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17100676
Record Dates: First submitted 2019-03-04; First posted 2019-03-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Spine Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLF (Active Comparator): posterolateral fusion
  Interventions: Procedure: posterolateral fusion
- PLIF (Active Comparator): posterior lumbar interbody fusion
  Interventions: Procedure: posterior lumbar interbody fusion

INTERVENTIONS:
Procedure: posterolateral fusion — Instrumented posterolateral fusion is a spinal surgery that combines bone graft fusion with the use of hardware like screws and rods to stabilize the spine, correct alignment, and promote successful fusion. It's used for various spinal conditions.
  Other Names: PLF
  Arms: PLF
Procedure: posterior lumbar interbody fusion — Posterior lumbar interbody fusion (PLIF) is a spinal surgery that involves removing problematic discs, inserting bone graft material, and sometimes a spacer, to promote fusion and stabilize the spine.
  Other Names: PLIF
  Arms: PLIF

SUMMARY:
To compare postoperative radiographic sagittal parameters after monosegmental lumbar fusion: posterior lumbar interbody fusion versus postrolateral fusion in treatment of lumbar spine instability

DETAILED DESCRIPTION:
The term "spondylolisthesis" refers to slipping of a vertebra relative to an adjacent vertebra,and there are two mean types degenerative and lytic : Degenerative spondylolisthesis is secondary to osteoarthritis leading to facet incompetence and disc degeneration.This condition allows anterior translation of one vertebra on another. Spondylolysis is the break in the pars interarticularis and is the precursor of lytic spondylolisthesis which associated with a pars fracture When nonoperative care fails and surgery is being considered, the type of fusion should be tailored to the specific pathology being treated.So there are different operations to correct this instability like postrolateral fusion (PLF) and posterior lumber interbody fusion (PLIF) PLF decreases segmental motion in the posterior column, which presumably reduces facet joint pain.Theoretical advantages of PLIF include decompression of exiting nerve roots by distraction of the collapsed disc space, achievement of optimal fusion in relation to the load-bearing capacity of the vertebral bodies and possibly attainment of a better fusion rate

ELIGIBILITY:
Inclusion Criteria:

* Adult patient older of 18 years old.
* Patients with lytic spondylolisthesis
* Low grade spondylolisthsis 1,2

Exclusion Criteria:

* Traumatic spondylolysis
* Previous spine surgery.
* Patient younger 18 years old
* High grade spondylolisthsis 3,4,5 - multiple levels spondylolithises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Spino sacral angle | 6month post op
  Which is the angle fromed between the line from front side of t1 to the middle of sacrum and the line passing through the sacral plateau

SECONDARY OUTCOMES:
T1 pelvic angle | Pre op. Post op immediately. 6month post op
  The angle between the line from centroid of t1 to the femoral head axis and the line from femoral head axis to middle of the s1 end plate
Pelvic incidence | Pre op. Post op immediately. 6month post op
  Is the angle between the line perpendicular to the s1 end plate from the midpoint of the end plate and the connecting line from the midpoint of the s1 end plate to center of the femoral head
Pelvic tilt | Pre op. Post op immediately. 6month post op
  Is the angle between the connecting line from the midpoint of the s1 end plate to the center of the femoral head and the vertical line
Sacral slope | Pre op. Post op immediately. 6month post op
  Is the angle between the tangent and the horizontal line of s1 end plate
Lumbar lordosis | Pre op. Post op immediately. 6month post op
  Is the junction of the thoracic kyphosis to the s1 end plate

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud fouad, lecturer, Study Director — assuit university hospitals
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

REFERENCES:
- [Background] Mobbs RJ, Phan K, Malham G, Seex K, Rao PJ. Lumbar interbody fusion: techniques, indications and comparison of interbody fusion options including PLIF, TLIF, MI-TLIF, OLIF/ATP, LLIF and ALIF. J Spine Surg. 2015 Dec;1(1):2-18. doi: 10.3978/j.issn.2414-469X.2015.10.05. PMID 27683674
- [Background] Madan S, Boeree NR. Outcome of posterior lumbar interbody fusion versus posterolateral fusion for spondylolytic spondylolisthesis. Spine (Phila Pa 1976). 2002 Jul 15;27(14):1536-42. doi: 10.1097/00007632-200207150-00011. PMID 12131714
- [Background] CLOWARD RB. The treatment of ruptured lumbar intervertebral discs by vertebral body fusion. I. Indications, operative technique, after care. J Neurosurg. 1953 Mar;10(2):154-68. doi: 10.3171/jns.1953.10.2.0154. No abstract available. PMID 13035484
- [Background] Cole CD, McCall TD, Schmidt MH, Dailey AT. Comparison of low back fusion techniques: transforaminal lumbar interbody fusion (TLIF) or posterior lumbar interbody fusion (PLIF) approaches. Curr Rev Musculoskelet Med. 2009 Jun;2(2):118-26. doi: 10.1007/s12178-009-9053-8. Epub 2009 Apr 29. PMID 19468868
- [Background] Kuraishi S, Takahashi J, Mukaiyama K, Shimizu M, Ikegami S, Futatsugi T, Hirabayashi H, Ogihara N, Hashidate H, Tateiwa Y, Kinoshita H, Kato H. Comparison of Clinical and Radiological Results of Posterolateral Fusion and Posterior Lumbar Interbody Fusion in the Treatment of L4 Degenerative Lumbar Spondylolisthesis. Asian Spine J. 2016 Feb;10(1):143-52. doi: 10.4184/asj.2016.10.1.143. Epub 2016 Feb 16. PMID 26949470
- [Background] Herkowitz HN, Kurz LT. Degenerative lumbar spondylolisthesis with spinal stenosis. A prospective study comparing decompression with decompression and intertransverse process arthrodesis. J Bone Joint Surg Am. 1991 Jul;73(6):802-8. PMID 2071615
- [Background] Feffer HL, Wiesel SW, Cuckler JM, Rothman RH. Degenerative spondylolisthesis. To fuse or not to fuse. Spine (Phila Pa 1976). 1985 Apr;10(3):287-9. PMID 3992350
- [Background] Lidar Z, Beaumont A, Lifshutz J, Maiman DJ. Clinical and radiological relationship between posterior lumbar interbody fusion and posterolateral lumbar fusion. Surg Neurol. 2005 Oct;64(4):303-8; discussion 308. doi: 10.1016/j.surneu.2005.03.025. PMID 16181997
- [Background] Hu SS, Tribus CB, Diab M, Ghanayem AJ. Spondylolisthesis and spondylolysis. J Bone Joint Surg Am. 2008 Mar;90(3):656-71. No abstract available. PMID 18326106